CLINICAL TRIAL: NCT02590913
Title: Acute Metabolic and Endocrine Responses of Glucose and Fructose in Healthy Young Subjects: A Double-blinded, Randomized, Crossover Trial
Brief Title: Acute Metabolic and Endocrine Responses of Glucose and Fructose in Healthy Young Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Duo li, Professor, Zhejiang University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: Zhejiang University
Record Dates: First submitted 2015-10-25; First posted 2015-10-29 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Healthy
Keywords: fructose; metabolism; acute
MeSH Terms: interventions — Fructose; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group fructose (Experimental): Volunteer was randomized into either group fructose or glucose
  Interventions: Dietary Supplement: fructose; Dietary Supplement: glucose
- group glucose (Experimental): After one-week washout period, volunteer was crossed over for either group glucose or fructose.
  Interventions: Dietary Supplement: fructose; Dietary Supplement: glucose

INTERVENTIONS:
Dietary Supplement: fructose — 75g fructose is dissolved in 300 ml water.After overnight fasting, 300ml of solution at 0830 within 5 minutes is taken by volunteers
Dietary Supplement: glucose — 75g glucose is dissolved in 300 ml water.After overnight fasting, 300ml of solution at 0830 within 5 minutes is taken by volunteers

SUMMARY:
The purpose of this study is to investigate the metabolic and endocrine responses during 3 hour after taking 75g fructose or glucose in young Chinese.

DETAILED DESCRIPTION:
The study was a double-blinded, randomized, crossover trial. Twenty healthy volunteers were randomized to two groups: group A (300ml of 22.5% glucose) and group B (300ml of 22.5% fructose).Volunteer was randomized into either group A or B, after an 8-h overnight fasting, took 300ml of solution at 0830 within 5 minutes. After one-week washout period, volunteer was crossed over for either group B or A. each intervention, venous blood was collected at 0h, 0.5h, 1h, 2h, and 3h and blood pressure was tested at 0h, 1h, 2h, and 3h.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were aged 19-39 years, with BMI between 18-24 kg/m 2.

Exclusion Criteria:

* Subjects pregnant or having a history of hepatic or renal disease, fructose intolerance, gout, hypoglycemia, or diabetes mellitus were excluded.
* Subjects taking any drugs, botanicals, or nutraceutical known to influence blood pressure also were rejected either.

Ages: 19 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
serum uric acid | 3 hours
  Serum uric acid concentration was analyzed on HITACHI 7020 chemistry analyzer using enzyme-based colorimetric test or colorimetric test supplied by DiaSys Diagnostic Systems (Shanghai) Co., Ltd

SECONDARY OUTCOMES:
blood pressure | 3 hours
  Blood pressure was measured at Zhejiang University Hospital by the research workers who were blind to the groups within 3 hours blood collection.

OTHER OUTCOMES:
serum glucose | 3 hours
  Serum glucose level was analyzed on HITACHI 7020 chemistry analyzer using enzyme-based colorimetric test or colorimetric test supplied by Diasys Diagnostic Systems (Shanghai) Co., Ltd
nitric oxide | 3 hours
  Serum nitric oxide concentration was measured using NO assay kit (Nanjing Jiancheng Technology Co., Lte., Nanjing, China) by the research workers who were blind to the groups.
aldose reductase | 3 hours
  Enzymatic activity of aldose reductase in serum was measured using ELISA kit (Shanghai Changjin Biology Co., Lte., Shanghai, China ) by the research workers who were blind to the groups.
phosphofructokinase | 3 hours
  Enzymatic activity of phosphofructokinase in serum was measured using ELISA kit (Shanghai Changjin Biology Co., Lte., Shanghai, China ) by the research workers who were blind to the groups .
insulin | 3 hours
  Serum insulin concentration was analyzed on HITACHI 7020 chemistry analyzer using enzyme-based colorimetric test or colorimetric test supplied by Diasys Diagnostic Systems (Shanghai) Co., Ltd
insulin-c | 3 hours
  Serum insulin-c concentration was analyzed on HITACHI 7020 chemistry analyzer using enzyme-based colorimetric test or colorimetric test supplied by Diasys Diagnostic Systems (Shanghai) Co., Ltd
triglyceride | 3 hours
  Triglyceride concentration in serum was analyzed on HITACHI 7020 chemistry analyzer using enzyme-based colorimetric test or colorimetric test supplied by Diasys Diagnostic Systems (Shanghai) Co., Ltd
total cholesterol | 3 hours
  Total cholesterol concentration was analyzed on HITACHI 7020 chemistry analyzer using enzyme-based colorimetric test or colorimetric test supplied by Diasys Diagnostic Systems (Shanghai) Co., Ltd
high-density cholesterol | 3 hours
  High-density cholesterol was analyzed on HITACHI 7020 chemistry analyzer using enzyme-based colorimetric test or colorimetric test supplied by Diasys Diagnostic Systems (Shanghai) Co., Ltd.
low-density cholesterol | 3 hours
  Low-density cholesterol concentration was analyzed on HITACHI 7020 chemistry analyzer using enzyme-based colorimetric test or colorimetric test supplied by Diasys Diagnostic Systems (Shanghai) Co., Ltd.
lactate dehydrogenase | 3 hours
  Enzymatic activity of lactate dehydrogenase was analyzed on HITACHI 7020 chemistry analyzer using enzyme-based colorimetric test or colorimetric test supplied by Diasys Diagnostic Systems (Shanghai) Co., Ltd.

CONTACTS AND LOCATIONS:
Overall Officials: Duo Li, Doctor, Study Director — College of Biosystem Engineering & Food Science, Zhejiang University
Locations (1):
- Zhejiang university, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Fulgoni V 3rd. High-fructose corn syrup: everything you wanted to know, but were afraid to ask. Am J Clin Nutr. 2008 Dec;88(6):1715S. doi: 10.3945/ajcn.2008.25825A. PMID 19064535
- [Background] Le MT, Frye RF, Rivard CJ, Cheng J, McFann KK, Segal MS, Johnson RJ, Johnson JA. Effects of high-fructose corn syrup and sucrose on the pharmacokinetics of fructose and acute metabolic and hemodynamic responses in healthy subjects. Metabolism. 2012 May;61(5):641-51. doi: 10.1016/j.metabol.2011.09.013. Epub 2011 Dec 5. PMID 22152650